CLINICAL TRIAL: NCT07260513
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of GH2616 in Subjects With Advanced Solid Tumor.
Acronym: GH2616C102
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Genhouse Bio Co., Ltd. (Other)
Collaborators: GCP ClinPlus Co., Ltd. (Unknown); Jiaxing Yidixi Computer Technology Co., Ltd (Unknown); Nanjing CR Medicon Technology Co., Ltd. (Unknown); Nanjing Shihejiyin Technology, Inc. (Industry); Fudan University (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GH2616C102
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GH2616 Tablet Group (Experimental): GH2616（Phase 1a：Dose Escalation） Subjects with advanced solid tumors harboring functional loss mutations of TP53 will be enrolled in dose escalation cohorts. Dose escalation of GH2616 will be conducted to determine the maximum tolerated dose (MTD).
  GH2616（Phase 1b：Dose Expansion） Depending on data obtained from the dose escalation part, dose expansion may proceed with multiple cohorts in subjects with advanced solid tumor harboring functional loss mutations of TP53 and whole genome doubling (WGD) characteristics.
  Interventions: Drug: GH2616 Tablets for oral administration at specified doses on scheduled days.

INTERVENTIONS:
Drug: GH2616 Tablets for oral administration at specified doses on scheduled days. — Drug: GH2616 Treatment group: Subjects will receive GH2616 orally in a dose escalation until confirmed progression, unacceptable toxicity, or any criterion for withdrawal from the study.

SUMMARY:
GH2616 is a potent and selective inhibitor targeting KIF18A, exhibiting distinct and superior anticancer properties compared to other cell cycle and anti-mitotic drug targets, with significant inhibitory effects on TP53 mutant and WGD (whole genome doubling) or CIN (chromosomal instability) tumors. GH2616 regulates chromosome distribution and alignment, prolongs mitotic duration, and activates the spindle assembly checkpoint by inhibiting KIF18A activity, thereby arresting mitosis at the G2/M phase, inducing mitotic catastrophe, and ultimately achieving tumor suppression.

This study will evaluate the safety and tolerability of GH2616 in patients with advanced solid tumors, and determine its dose-limiting toxicity (DLT), maximum tolerated dose (MTD), and/or recommended phase II dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

- 1.Female, aged ≥18 years. 2.Assessed by the investigator as suitable for participation in this study in the following two aspects: a. The subject fully understands the requirements of this study and voluntarily signs a written informed consent form; b. Can comply with the medication requirements of this study and all study-related procedures and assessments.

3.Tumor types meeting the following conditions:

Phase Ia:

Subjects with relapsed or metastatic advanced gynecological tumors and triple-negative breast cancer (TNBC) confirmed by histology or cytology and laboratory-confirmed functional loss mutation of TP53, including but not limited to high-grade serous ovarian cancer (HGSOC), uterine carcinosarcoma (UCS), endometrial cancer (EC) and other gynecological tumors, and TNBC.

Phase Ib:

Subjects with relapsed or metastatic advanced gynecological tumors and TNBC confirmed by histology or cytology and laboratory-confirmed functional loss mutation of TP53 and genomic doubling (WGD) characteristics, including but not limited to HGSOC, UCS, EC and other gynecological tumors, and TNBC. Specific requirements for each tumor type are as follows:

1. High-grade serous ovarian cancer: Platinum-resistant ovarian cancer that has progressed/relapsed after at least one line of platinum-containing chemotherapy, or platinum-sensitive ovarian cancer that has progressed/relapsed after at least two lines of platinum-containing chemotherapy. The definition of "platinum-resistant" is: the interval between the discovery of tumor recurrence and the last chemotherapy of the previous platinum-containing regimen is <6 months, or the tumor progresses during initial treatment or recurrence treatment. The definition of "platinum-sensitive" is: the interval between the discovery of tumor recurrence and the last chemotherapy is ≥6 months. The interval should be calculated from the date of the last platinum drug treatment to the date of disease progression.
2. Uterine carcinosarcoma: Progressed/relapsed after at least one line of platinum-containing chemotherapy.
3. Endometrial cancer: Progressed/relapsed after at least one line of platinum-containing chemotherapy.
4. TNBC: Progressed/relapsed after at least one line of chemotherapy. Note: Subjects receiving adjuvant therapy who have disease progression within less than 6 months after the end of treatment can be considered as having received first-line therapy.

4.Expected survival time ≥ 12 weeks. 5.Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1. 6.According to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 there is at least 1 measurable lesion. Lesions previously treated with local therapy such as radiotherapy are not considered measurable lesions unless there is definite progression after local therapy.

7.Subjects have sufficient vital organ function at screening (requirement: no blood transfusion, no use of hematopoietic stimulators or human albumin preparations within 14 days before screening), specifically defined as follows:

1. Blood routine: Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L; Platelet count (PLT) ≥100 × 10⁹/L or greater than the laboratory normal value; Hemoglobin (HGB) ≥90 g/L (9 g/dL).
2. Liver function: Serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN). For subjects with liver metastasis or confirmed Gilbert syndrome, TBIL ≤ 3 × ULN. For subjects without liver metastasis, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN. For subjects with liver metastasis, ALT or AST ≤ 5 × ULN.
3. Renal function: Creatinine clearance (CLCr) calculated by the Cockcroft-Gault method (Appendix 3: Creatinine Clearance Calculation Formula) ≥ 60 mL/min.
4. Coagulation function: Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤ 2 × ULN (indicators of subjects receiving anticoagulant therapy are within the therapeutic range).
5. Cardiac function standard: Echocardiogram (ECHO) shows left ventricular ejection fraction greater than 50%.

   8.Serum pregnancy test of female subjects of childbearing age within 7 days before the first use of the study drug must be negative; eligible subjects with fertility must agree to use reliable contraceptive methods (hormonal or barrier methods or abstinence, etc.) with their partners during the trial and for at least 3 months after the last dose. A subject with fertility is defined as sexually mature and having biological potential fertility.

Exclusion Criteria:

* 1.Received chemotherapy within 21 days before the first administration of GH2616 tablets, or received radiotherapy, endocrine therapy, immunotherapy and other anti-tumor drug treatments within 28 days before, and special regulations are made for the following anti-tumor drugs or treatments:

  1. Nitrosourea or mitomycin C: within 6 weeks before the first use of the study drug;
  2. Oral fluoropyrimidines, small molecule targeted drugs, and traditional Chinese medicine with anti-tumor indications: within 5 half-lives or 14 days before the first use of the study drug (whichever is shorter);
  3. Local palliative radiotherapy: within 14 days before the first use of the study drug.

  2.Received other unmarketed clinical research drugs or treatments within 28 days before the first administration.

  3.Acute toxicity caused by previous anti-tumor treatment before the first administration has not recovered to ≤ Grade 1 of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 or the baseline level specified in the inclusion criteria (except for toxicity such as alopecia and fatigue that the investigator judges to have no safety risk).

  4.Mean corrected QT interval (QTc, using Fridericia's correction formula) > 470 ms in resting 12-lead electrocardiogram (ECG) examination (ECG testing frequency can be increased if there are clinical indications). Various clinically significant arrhythmias, conduction, and resting ECG morphological abnormalities, such as complete left bundle branch block, third-degree heart block, etc. Various factors that may increase the risk of QTc prolongation or arrhythmic events, such as Class III heart failure, refractory hypokalemia, congenital long QT syndrome, and first-degree relatives with long QT syndrome in the family history.

  5.Have persistent or active infection, including: Active hepatitis B (hepatitis B surface antigen (HbsAg) positive and hepatitis B virus deoxyribonucleic acid (HBV-DNA) > 1000 IU/ml or 2000 cps/ml]; Patients infected with hepatitis C virus (defined as positive HCV antibody and HCV-RNA > upper limit of normal).

  6.Symptomatic or active progressive central nervous system (CNS) metastasis. 7.Uncontrolled concurrent diseases, such as:
  1. Severe infection within 14 days before starting study treatment, including but not limited to hospitalization for infection, bacteremia, or severe pneumonia complications; or received therapeutic intravenous antibiotics within two weeks before starting study treatment. Subjects using prophylactic antibiotics for biopsy can be enrolled;
  2. Heart failure meeting New York Heart Association functional class ≥III within 6 months before starting study treatment;
  3. Having other malignant tumors within 5 years before starting treatment or at the same time (except for in situ cancers such as non-melanoma skin basal cell carcinoma or squamous cell carcinoma, breast/cervical carcinoma in situ, superficial bladder cancer, etc. that have been radically treated and have no evidence of disease recurrence);
  4. Subjects with current or previous history of carcinomatous meningitis, spinal cord compression, etc.;
  5. Uncontrolled hypertension within 7 days before starting study treatment, defined as systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg even under treatment with multiple antihypertensive drugs;
  6. Any arterial thromboembolic event within 6 months before starting study treatment, including acute myocardial infarction, cerebrovascular accident, or transient ischemic attack;
  7. Tumor invades surrounding vital organs or blood vessels (such as mediastinal great vessels, superior vena cava, trachea, esophagus, etc.), or there is a risk of developing esophagotracheal fistula or esophagopleural fistula;
  8. After esophageal or tracheal lumen stent implantation;
  9. History of gastrointestinal perforation and/or fistula within 6 months before starting study treatment;
  10. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (once a month or more frequently);
  11. Uncontrolled tumor-related pain, or no stable pain treatment plan. 8.Allergic to GH2616 tablets or its formulation components. 9.Have significant impact on oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction.

      10.Subjects have severe underlying lung disease or history, such as severe chronic obstructive pulmonary disease, unhealed interstitial lung disease, unhealed acute or chronic infectious pneumonia, lung transplantation, etc.

      11.Use of strong inhibitors and strong inducers of P-glycoprotein (P-gp) within 14 days or 5 half-lives before the first administration (whichever is longer).

      12.Pregnant or lactating women. 13.Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.

      14.Underwent major surgical operations (craniotomy, thoracotomy, laparotomy, vascular interventional surgery) within 28 days before the first administration, or have unhealed wounds, ulcers, or fractures. Note: Local surgical treatment for isolated lesions for palliative purposes is acceptable.

      15.Previous history of definite mental disorder and taking medication for treatment.

      16.Previous treatment with KIF18A inhibitor. 17.Have POLE hotspot mutation, dMMR/MSI-H, or identifiable hypermutator phenotype.

      18.The investigator deems that the subject is not suitable to participate in this clinical study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) (according to NCI CTCAE 5.0). | From the initiation of study treatment to the completion of safety follow-up after the end of study treatment. Approximately 2 years.
  Evaluated at each dose level GH2616, as graded by National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) version 5.0.
Phase Ia: Dose Limited Toxicity (DLT) | 21 Days (first cycle)
  Evaluated at each dose level GH2616, as graded by National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) version 5.0.
Phase Ib: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) (according to NCI CTCAE 5.0). | From the initiation of study treatment to the completion of safety follow-up after the end of study treatment. Approximately 2 years.
  Evaluated at each dose level GH2616, as graded by National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) version 5.0.
Phase Ib:- Objective response rate (ORR) | Day 1 through 12 cycles (each cycle is 21 days)
  The number (%) of patients with a best overall response of complete response (CR) or partial response (PR) per RECIST v1.1 as assessed by investigator.

SECONDARY OUTCOMES:
Phase Ia and Phase Ib-- Evaluation of pharmacokinetics: plasma concentrations at different times after dosing and related assessment of conventional pharmacokinetic parameters | From the initiation of study treatment to the completion of safety follow-up after the end of study treatment.
Phase Ia and Phase Ib--Duration of Response (DOR) | From the initiation of study treatment to the completion of safety follow-up after the end of study treatment.
  Antitumor activity was evaluated by assessing tumor response using RECIST 1.1 criteria.
Phase Ia and Phase Ib--Disease Control Rate (DCR) | From the initiation of study treatment to the completion of safety follow-up after the end of study treatment.
  Antitumor activity was evaluated by assessing tumor response using RECIST 1.1 criteria.
Phase Ia and Phase Ib--Progression-Free Survival (PFS) | From the initiation of study treatment to the completion of safety follow-up after the end of study treatment.
  Antitumor activity was evaluated by assessing tumor response using RECIST 1.1 criteria.
Phase Ib--Overall Survival (OS) | From the initiation of study treatment to the completion of safety follow-up after the end of study treatment.
  Antitumor activity was evaluated by assessing tumor response using RECIST 1.1 criteria.
Phase Ia and Phase Ib--QT Interval Evaluation. | Collection will be conducted until Cycle 13.
  To assess the relationship between plasma concentrations of GH2616 Tablets and QT interval changes in subjects with advanced solid tumors after oral administration.

CONTACTS AND LOCATIONS:
Overall Officials: QIAN DONG, MASTER, Study Director — Suzhou Genhouse Bio Co., Ltd.
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No